CLINICAL TRIAL: NCT03489265
Title: Treatment of Diarrhea-Associated Fecal Incontinence With Eluxadoline
Brief Title: Effects of Eluxadoline (Viberzi®) 100 mg Twice Daily on Diarrhea-Associated Fecal Incontinence
Acronym: ELXDFI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult to recruit severely affected patients with fecal incontinence
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-1561; 895 (Other Grant/Funding Number: Allergan Pharmaceutical)
Record Dates: First submitted 2018-03-09; First posted 2018-04-05 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Fecal Incontinence; Accidental Bowel Leakage; Anal Incontinence; Diarrhea; Urge Incontinence
MeSH Terms: conditions — Fecal Incontinence; Encopresis; Diarrhea; Urinary Incontinence, Urge | interventions — eluxadoline; Sugars

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 1 of 2 sequences. Each sequence includes 4 periods: Run-in, Treatment Period 1, Treatment Period 2, and Follow-Up. In Sequence A, Eluxadoline will be given 100 mg BID in Treatment Period 1 and Placebo will be given in Treatment Period 2. In Sequence B, Placebo will be given in Treatment Period 1 and Eluxadoline will be given in Treatment Period 2. Placebo will be given during Baseline and Follow-Up of both arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will not be aware when Eluxadoline or Placebo are administered. Investigators will be masked to whether Eluxadoline is given in Treatment Period 1 or Treatment Period 2 unless there is an adverse event that requires unmasking the treatment for this patient to ascertain whether the adverse event is drug-related.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eluxadoline followed by Placebo (Other): Following a 2-week run-in period, patients will receive Eluxadoline 100 mg twice daily for 4 weeks then placebo tablets taken twice daily for 4 weeks followed by a 2-week follow-up period during which placebo will be administered twice daily.
  Interventions: Drug: Eluxadoline 100 mg; Other: Placebo
- Placebo followed by Eluxadoline (Other): Following a 2-week run-in period, patients will receive placebo twice daily for 4 weeks then Eluxadoline 100 mg twice daily for 4 weeks followed by a 2-week follow-up period during which placebo will be administered twice daily.
  Interventions: Drug: Eluxadoline 100 mg; Other: Placebo

INTERVENTIONS:
Drug: Eluxadoline 100 mg — 100 mg capsule-shaped tablet by mouth taken twice per day
  Other Names: Viberzi®
Other: Placebo — Matching capsule-shaped placebo tablets taken by mouth twice per day
  Other Names: sugar pill

SUMMARY:
Accidental bowel leakage (fecal incontinence) increases in people who have diarrhea and sensations of urgency to have a bowel movement. Drugs such as loperamide (Imodium) that reduce diarrhea improve accidental bowel leakage, but loperamide has disadvantages: it is difficult to find a dose that does not cause constipation, and it does not reduce urge sensations. Eluxadoline is a new drug that is effective for reducing diarrhea, abdominal pain, and urgency in patients with irritable bowel syndrome, and it may be less likely than loperamide to cause severe constipation. Therefore, eluxadoline may help patients manage accidental bowel leakage caused by diarrhea. The chemical name for Viberzi® is eluxadoline.

The primary aims of this study are to find out if eluxadoline at a dose of 100 mg orally twice a day will reduce the average number of days the patient has accidental bowel leakage, and to see if the rate of accidental bowel leakage increases when the patient stops taking eluxadoline. Additional goals are to find out if eluxadoline decreases diarrhea and urge sensations.

This is a small (pilot) study to show whether eluxadoline is an effective way of treating accidental bowel leakage. If the study shows this, a larger study will be needed. There are three phases to this 12-week study: (1) A two-week run-in period to see if the patient meets the inclusion criteria. (2) Two months for treatment including one month on eluxadoline and one on placebo (sugar pills) twice a day. (3) A two-week follow-up to see what happens when you stop taking eluxadoline.

To participate in the study, patients should be aged 18 or older. Patients with inflammatory bowel disease, anal fissures, or congenital malformations will be excluded.

The primary outcome is the average number of days per week with any solid or liquid bowel accidents. Additional information includes: (1) Number of days per week the patient takes loperamide, (2) days per week with loose or watery stools, (3) days per week with moderate to strong urge sensations, and (4) questionnaires to measure the severity of accidental bowel leakage, quality of life, anxiety, and depression. There will be up to 38 patients in the study.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Any gender, race, or ethnicity.
3. Must self-report an average of at least 2 episodes of solid or liquid FI per week for the previous month.
4. Must self-report an average of at least 2 bowel movements (BMs) per week that are Bristol Types 6 or 7 (mushy or liquid stools).
5. Subjects must have access to the internet at home and be willing to enter symptom data each night before sleeping.

Exclusion Criteria:

1. Patients with inflammatory bowel disease, anal fissure, or congenital malformations as a cause of FI will be excluded.
2. Subjects who start the study and do not experience at least 4 episodes of solid or liquid FI and at least 4 BMs that are Bristol Stool types 6 or 7 during the first two weeks will be withdrawn from the study.
3. Subjects who do not provide at least 4 days of valid stool diary data per week during the first two weeks will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Run-in days per week with fecal incontinence | Baseline Period, starting on Day 1 and ending at the conclusion of Day 14
  If there are less than 5 days in a 7-day period that have complete diary data, the subject will be excluded. The number of days per week with fecal incontinence (i.e., a score >0) will be counted and divided by 7 to obtain a rate per week. The range of scores is 0 to 7 with 7 being the most severe fecal incontinence.
Treatment Period 1 days per week with fecal incontinence | Treatment Period 1 (measured across Weeks 5 and 6)
  If there are less than 5 days in a 7-day period that have complete diary data in weeks 5 and 6, the Treatment Period 1 variable will be missing. The number of days per week with fecal incontinence (i.e., a score >0) will be counted and divided by 7 to obtain a rate per week. The range of scores is 0 to 7 with 7 being the most severe fecal incontinence.
Treatment Period 2 days per week with fecal incontinence | Treatment Period 2 (measured across Weeks 9 and 10)
  If there are less than 5 days in a 7-day period that have complete diary data in weeks 9 and 10, the Treatment Period 2 variable is missing. The number of days per week with fecal incontinence (i.e., a score >0) will be counted and divided by 7 to obtain a rate per week. The range of scores is 0 to 7 with 7 being the most severe fecal incontinence.
Follow-up days per week with fecal incontinence | Follow-up period (measured across Weeks 11 and 12)
  If there are less than 5 days in a 7-day period that have complete diary data in weeks 11 and 12, the Follow-Up variable is missing. The number of days per week with fecal incontinence (i.e., a score >0) will be counted and divided by 7 to obtain a rate per week. The range of scores is 0 to 7 with 7 being the most severe fecal incontinence.

SECONDARY OUTCOMES:
Days per week with loperamide (escape medication) | Weeks 1, 2, 5, 6, 9, 10, 11, and 12
  For eligibility analysis, Run-in (Weeks 1 and 2) will determine if there are 5 to 7 days in each week that can be evaluated; if less than one week, the subject is excluded. For treatment assessment, Treatment Period 1 (Weeks 5 and 6) and Treatment Period 2 (Weeks 9 and 10) will determine if there are 5 to 7 days that can be evaluated; if less than one week per period, the subject will be excluded from analysis. For evaluation of drug withdrawal, Follow-up (Weeks 11 and 12) will be examined to determine if there are 5 to 7 days that can be evaluated; if less than one week, the data is missing. In all analyses, count the number of days in each period with any loperamide used. The range of scores is 0 to 7 with 7 being the greatest amount of rescue medication used.
Days per week patient described bowel movements as 6 or 7 on the Bristol Stool Scale | Weeks 1, 2, 5, 6, 9, 10, 11, and 12
  For eligibility analysis, Run-in (Weeks 1 and 2) will determine if there are 5 to 7 days in each week that can be evaluated; if less than one week, the subject is excluded. For treatment assessment, Treatment Period 1 (Weeks 5 and 6) and Treatment Period 2 (Weeks 9 and 10) will determine if there are 5 to 7 days that can be evaluated; if less than one week per period, the subject will be excluded from analysis. For evaluation of drug withdrawal, Follow-up (Weeks 11 and 12) will be examined to determine if there are 5 to 7 days that can be evaluated; if less than one week, the data is missing. In all analyses, count the number of days in each period with any Bristol Stool Scale score of 6 or 7. The range of scores is 0 to 7 days with 7 being the most severe diarrhea.
Days per week patient reported strong urge sensations | Weeks 1, 2, 5, 6, 9, 10, 11, and 12
  For eligibility analysis, Run-in (Weeks 1 and 2) will determine if there are 5 to 7 days in each week that can be evaluated; if less than one week, the subject is excluded. For treatment assessment, Treatment Period 1 (Weeks 5 and 6) and Treatment Period 2 (Weeks 9 and 10) will determine if there are 5 to 7 days that can be evaluated; if less than one week per period, the subject will be excluded from analysis. For evaluation of drug withdrawal, Follow-up (Weeks 11 and 12) will be examined to determine if there are 5 to 7 days that can be evaluated; if less than one week, the data is missing. In all analyses, count the number of days in each period with any moderate to strong urge sensations . The range of scores is 0 to 7 days with 7 being the most severe urgency to defecate.
Fecal Incontinence Severity Score (FISS) over time | Weeks 2, 6,10, and 12
  For clinic visits in Weeks 2, 6, 10, and 12, compute the score for the 4 components of the FISS. These components are frequency of leaks, type of leakage, amount that leaked, and urgency vs. passive incontinence. These individual items are added together to form a total score which ranges from 3 to 13, with 13 representing the most severe form of fecal incontinence (FI). If items are not completed or are not correct, the FISS score is missing.
Fecal Incontinence Quality of Life Scale Score for Lifestyle (FIQOL-Lifestyle) | Weeks 2, 6, 10, and12
  For clinic visits in Weeks 2, 6, 10, and 12, compute the scale score for lifestyle. If more than half of the items in the scale are present, the score is based on the average for those items; otherwise the FIQOL-Lifestyle scale score is missing. Scores range from 0 to 4 with 4 representing the greatest impairment in FIQOL-Lifestyle.
Fecal Incontinence Quality of Life Scale Score for Coping/Behavior (FIQOL-Coping/Behavior) | Weeks 2, 6, 10, and 12
  For clinic visits in Weeks 2, 6, 10, and 12, compute the scale score for Coping/Behavior. If more than half of the items in the scale are present, the score is based on the average for those items; otherwise the FIQOL-Coping/Behavior scale score is missing. Scores range from 0 to 4 with 4 representing the greatest impairment in FIQOL-Coping/Behavior.
Fecal Incontinence Quality of Life Scale Score for Depression/Self-Perception (FIQOL-Depression/Self-Perception) | Weeks 2, 6, 10, and 12
  For clinic visits in Weeks 2, 6, 10, and 12, compute the scale score for Depression/Self-Perception. If more than half of the items in the scale are present, the score is based on the average for those items; otherwise the FIQOL-Depression/Self-Perception scale score is missing. Scores range from 0 to 4 with 4 representing the greatest impairment in FIQOL-Depression/Self-Perception.
Fecal Incontinence Quality of Life Scale Score for Embarrassment (FIQOL-Embarrassment) | Weeks 2, 6, 10, and 12
  For clinic visits in Weeks 2, 6, 10, and 12, compute the scale score for Embarrassment. If more than half of the items in the scale are present, the score is based on the average for those items; otherwise the FIQOL-Embarrassment scale score is missing. Scores range from 0 to 4 with 4 representing the greatest impairment in FIQOL-Embarrassment.
Brief Symptom Inventory-18 Anxiety Score (BSI-Anxiety) | Weeks 2, 6, 10, and 12
  For each visit to the clinic, compute the previous week's BSI scores for anxiety. If more than two items are not answered, the score is not valid. Scores of 0 to 4 are added across items with missing items being replaced by the average for the present items, and the summary score is transformed into a T-score in which the average score is 50 and 10 is equivalent to a standard deviation in the reference sample. A score of 60 represents one standard deviation above the population mean for severity of anxiety.
Brief Symptom Inventory-18 Depression Score (BSI-Depression) | Weeks 2, 6, 10, and 12
  For each visit to the clinic, compute the previous week's BSI scores for depression. If more than two items are not answered, the score is not valid. Scores of 0 to 4 are added across items with missing items being replaced by the average for the present items, and the summary score is transformed into a T-score in which the average score is 50 and 10 is equivalent to a standard deviation in the reference sample. A score of 60 represents one standard deviation above the population mean for severity of depression.
Preference for study drug vs. loperamide | Weeks 6, and 10
  On Week 6 and 10, subject will be asked to compare the study drug to loperamide for the previous 4 weeks. The choices are -2=strongly prefer loperamide, -1=somewhat prefer loperamide, 0=no preference, 1=somewhat prefer study drug, and 2=strongly prefer study drug. The range of scores is -2 to +2, with +2 being equivalent to a strong preference for the study drug over loperamide.
Preference for eluxadoline or placebo | Week 10
  At week 10, subjects will be asked to compare the second study drug to the first study drug for the previous 8 weeks. For subjects randomized to the "Eluxadoline followed by Placebo" group, the first study drug is eluxadoline; for subjects in the "Placebo followed by Eluxadoline" group the second study drug is eluxadoline. To estimate the preference of subjects for eluxadoline, the preference of the first group for the first study period and the preferences of the second group for the second study period will be averaged. The range of outcome scores is -2 to +2 with +2 representing a strong preference for eluxadoline over placebo. (The excluded groups are available as a way to assess whether order effects interfere with the measurement of preferences for eluxadoline vs. placebo.)

CONTACTS AND LOCATIONS:
Overall Officials: William (Bill) Whitehead, PhD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB) and executes a data use/sharing agreement with the University of North Carolina.
Supporting Information: CSR, Analytic Code
Time Frame: 9-36 months following publication of the study results.
Access Criteria: Requester must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IED), or Research Ethics Board (REB), and requester has executed an acceptable data use/sharing agreement with UNC.
URL: https://irbis2.research.unc.edu/irb/

REFERENCES:
- [Background] Whitehead WE, Borrud L, Goode PS, Meikle S, Mueller ER, Tuteja A, Weidner A, Weinstein M, Ye W; Pelvic Floor Disorders Network. Fecal incontinence in US adults: epidemiology and risk factors. Gastroenterology. 2009 Aug;137(2):512-7, 517.e1-2. doi: 10.1053/j.gastro.2009.04.054. Epub 2009 May 4. PMID 19410574
- [Background] Bharucha AE, Zinsmeister AR, Locke GR, Seide BM, McKeon K, Schleck CD, Melton LJ 3rd. Risk factors for fecal incontinence: a population-based study in women. Am J Gastroenterol. 2006 Jun;101(6):1305-12. doi: 10.1111/j.1572-0241.2006.00553.x. PMID 16771954
- [Background] Lembo AJ, Lacy BE, Zuckerman MJ, Schey R, Dove LS, Andrae DA, Davenport JM, McIntyre G, Lopez R, Turner L, Covington PS. Eluxadoline for Irritable Bowel Syndrome with Diarrhea. N Engl J Med. 2016 Jan 21;374(3):242-53. doi: 10.1056/NEJMoa1505180. PMID 26789872
- [Background] Simren M, Palsson OS, Heymen S, Bajor A, Tornblom H, Whitehead WE. Fecal incontinence in irritable bowel syndrome: Prevalence and associated factors in Swedish and American patients. Neurogastroenterol Motil. 2017 Feb;29(2):10.1111/nmo.12919. doi: 10.1111/nmo.12919. Epub 2016 Aug 31. PMID 27581702
- [Background] Sun WM, Read NW, Verlinden M. Effects of loperamide oxide on gastrointestinal transit time and anorectal function in patients with chronic diarrhoea and faecal incontinence. Scand J Gastroenterol. 1997 Jan;32(1):34-8. doi: 10.3109/00365529709025060. PMID 9018764
- [Background] Sjodahl J, Walter SA, Johansson E, Ingemansson A, Ryn AK, Hallbook O. Combination therapy with biofeedback, loperamide, and stool-bulking agents is effective for the treatment of fecal incontinence in women - a randomized controlled trial. Scand J Gastroenterol. 2015 Aug;50(8):965-74. doi: 10.3109/00365521.2014.999252. Epub 2015 Apr 20. PMID 25892434
- [Background] Palmer KR, Corbett CL, Holdsworth CD. Double-blind cross-over study comparing loperamide, codeine and diphenoxylate in the treatment of chronic diarrhea. Gastroenterology. 1980 Dec;79(6):1272-5. PMID 7002706
- [Background] Dove LS, Lembo A, Randall CW, Fogel R, Andrae D, Davenport JM, McIntyre G, Almenoff JS, Covington PS. Eluxadoline benefits patients with irritable bowel syndrome with diarrhea in a phase 2 study. Gastroenterology. 2013 Aug;145(2):329-38.e1. doi: 10.1053/j.gastro.2013.04.006. Epub 2013 Apr 9. PMID 23583433
- [Background] Noelting J, Zinsmeister AR, Bharucha AE. Validating endpoints for therapeutic trials in fecal incontinence. Neurogastroenterol Motil. 2016 Aug;28(8):1148-56. doi: 10.1111/nmo.12809. Epub 2016 Mar 6. PMID 26948292
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117
- [Background] Read M, Read NW, Barber DC, Duthie HL. Effects of loperamide on anal sphincter function in patients complaining of chronic diarrhea with fecal incontinence and urgency. Dig Dis Sci. 1982 Sep;27(9):807-14. doi: 10.1007/BF01391374. PMID 7105952
- See also: Link to Eluxadoline (Viberzi) Patient Information Guide and full prescribing information provided by Allergan — http://www.allergan.com/assets/pdf/viberzi_pi